CLINICAL TRIAL: NCT05845294
Title: A Study of the Effect of Short-term Structured Psychological Care on the Level of Postoperative Stigma in Patients With Colorectal Cancer
Brief Title: A Study of the Effect of Short-term Structured Psychological Care in Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zunyi Medical College (Other)
Responsible Party: Principal Investigator, Xu Ren, Study Director, Zunyi Medical College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Zunyi002
Record Dates: First submitted 2023-04-13; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator)
  Interventions: Procedure: Routine Care
- Experimental group (Experimental)
  Interventions: Procedure: Short-term structured psychological Care

INTERVENTIONS:
Procedure: Routine Care — Routine care for patients undergoing colorectal cancer stoma
  Arms: Control group
Procedure: Short-term structured psychological Care — Short-term structured psychological care for colorectal cancer stoma patients based on conventional care
  Arms: Experimental group

SUMMARY:
The study explored the effects of short-term structured psychological care on the level of postoperative psychological resilience, stigma, anxiety and depression in patients with colorectal cancer colostomy.

ELIGIBILITY:
Inclusion Criteria:

1. voluntary participation in the study and ability to cooperate with treatment and care;
2. patients who were to undergo enterostomy;
3. age ≥18 years;
4. consciousness (being able to complete the questionnaire alone or able to answer the questions correctly);
5. social impact scale (SIS) score ≥24.

Exclusion Criteria:

1. Critically ill and unable to cooperate with the study;
2. Impaired cognitive function that affects communication;
3. Patients with other organic diseases in combination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Anxiety of patients was assessed by Chinese version of the Mental Toughness Scale | 1 month
  Anxiety of patients was assessed by Chinese version of the Mental Toughness Scale
Anxiety of patients was assessed by the Social Impact Scale | 1 month
  Anxiety of patients was assessed by the Social Impact Scale
Anxiety of patients was assessed by Hospital Anxiety and Depression Scale | 1 month
  Anxiety of patients was assessed by Hospital Anxiety and Depression Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Zunyi Medical College, Zunyi, Guizhou, China